CLINICAL TRIAL: NCT00053014
Title: S0125, A Phase II Study Of Chimerism-Mediated Immunotherapy (CMI) Using Nonmyeloablative Allogeneic Peripheral Blood Stem Cell Transplantation In Older Patients With Acute Myeloid Leukemia (AML) In First Complete Remission (A BMT Study)
Brief Title: S0125, Chemotherapy, Total-Body Irradiation, and Peripheral Stem Cell Transplantation in Treating Older Patients With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0125; S0125 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia in remission; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities
MeSH Terms: conditions — Leukemia; Congenital Abnormalities | interventions — Cyclosporine; fludarabine; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): patient conditioning - fludarabine 30 mg/m2 IV over 1 hour Days -4, -3, -2; TBI 6-7 cGy/min Day 0 post-transplant immunosuppression - cyclosporine 6.25 mg/kg bid PO D -3 to +180 (begin taper on D+35); mycophenolate mofetil 15mg/kg bid PO D0 to +27
  Interventions: Biological: therapeutic allogeneic lymphocytes; Drug: cyclosporine; Drug: fludarabine; Drug: mycophenolate mofetil; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes
Drug: cyclosporine
Drug: fludarabine
Drug: mycophenolate mofetil
  Other Names: MMF
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy and radiation therapy. Sometimes the transplanted cells can make an immune response against the body's normal tissues. Cyclosporine and mycophenolate mofetil may prevent this from happening.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy and total-body irradiation followed by donor peripheral stem cell transplantation, cyclosporine, and mycophenolate mofetil in treating older patients who have acute myeloid leukemia.

DETAILED DESCRIPTION:
Primary objective:

* Determine whether allogeneic peripheral blood stem cell transplantation with pre-conditioning low dose total body irradiation and fludarabine followed by cyclosporine and mycophenolate mofetil, when given to elderly patients with acute myeloid leukemia in first complete remission, is sufficiently efficacious (in terms of survival 1 year after transplantation) to warrant a phase III investigation.

Secondary objective:

* Determine the frequency and severity of toxic effects of this regimen in these patients.

Other objectives as funding permits:

* Determine whether chimerism patterns in bone marrow and blood after transplantation are associated with relapse and/or graft-versus-host disease (GVHD) in these patients.
* Determine whether cytogenic, immunophenotypic, and molecular biologic features detected in pre- and post-transplantation specimens are related to transplant outcomes and risk of relapse in these patients.

OUTLINE: This is an open-label study.

* Conditioning regimen: Patients receive fludarabine IV over 1 hour on days -4 to -2. Patients also undergo total body irradiation on day 0.
* Peripheral blood stem cell infusion (PBSC): Patients receive unmodified filgrastim transplantation (G-CSF)-mobilized donor PBSC on day 0.
* Post-transplantation immunosuppression: Patients receive oral cyclosporine on days -3 to 35 followed by a taper until day 180. Patients also receive oral mycophenolate mofetil on day 0 to 27 without tapering.
* Donor lymphocyte infusions (DLI): Patients with relapsed disease receive DLI IV over 30 minutes for up to 2 infusions.

Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 25-51 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologically confirmed acute myeloid leukemia (AML) (within 180 days of diagnosis) OR
* Secondary AML (secondary to myelodysplastic syndromes (MDS) or to prior leukemogenic therapy)
* Must have A1 marrow, B1 blood, and C1 extramedullary disease status
* Must have received prior remission induction chemotherapy
* Must have a genotypically HLA-identical sibling donor available that is not a monozygotic identical twin
* No M3 AML or blastic transformation of chronic myelogenous leukemia
* If history of CNS leukemia, no leukemia cells in CNS by lumbar puncture within past 7 days
* Must be concurrently enrolled on protocols SWOG-9007 and SWOG-S9910

PATIENT CHARACTERISTICS:

Age

* 55 to 69

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No other malignancy within the past 2 years except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Adequately treated stage I or II cancer in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior allogeneic hematopoietic stem cell transplantation

Chemotherapy

* See Disease Characteristics
* Prior consolidation therapy allowed

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Prior organ transplantation allowed provided not concurrently receiving immunosuppressive therapy

Ages: 55 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2003-04; Primary Completion 2005-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter McSweeney, MD, Study Chair — Rocky Mountain Cancer Centers - Denver Midtown
Locations (83):
- United States (83):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Scripps Cancer Center at Scripps Clinic, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - General Robert Huyser Cancer Center at David Grant Medical Center, Travis Air Force Base, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Mountain States Tumor Institute - Boise, Boise, Idaho
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Indiana Blood and Marrow Transplantation, Beech Grove, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - New Orleans Cancer Institute at Memorial Medical Center, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - University of Tennessee Cancer Institute at Methodist Central Hospital, Memphis, Tennessee
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Baylor College of Medicine, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: patient conditioning - fludarabine 30 mg/m2 IV over 1 hour Days -4, -3, -2; TBI 6-7 cGy/min Day 0 post-transplant immunosuppression - CSP 6.25 mg/kg bid PO D -3 to +180 (begin taper on D+35); MMF 15mg/kg bid PO D0 to +27
Period: Overall Study
Arm/Group | Treatment
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 62 [56 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: measured from date of registration to study until death from any cause with patients still alive censored at date of last contact
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
participants | 1

2. Secondary Outcome: Serious Adverse Events
Description: Twice a week for the first two months, one time a week during month 3, one time every two weeks for months 4-9.
Time Frame: 9 months
Population: All patients
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
participants | 0

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=5)
Infection and dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No